CLINICAL TRIAL: NCT02604732
Title: Randomized Controlled Trial on Pre-operative Withdrawal Versus no Withdrawal of Aspirin in Laparoscopic Inguinal Hernia Repair
Brief Title: Pre-operative Withdrawal of Aspirin in Laparoscopic Inguinal Hernia Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2015/00512
Record Dates: First submitted 2015-11-10; First posted 2015-11-13 (Estimated); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Inguinal Hernia
Keywords: Inguinal Hernia; Laparoscopic Inguinal Hernia Repair; Aspirin
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients who stop Aspirin perioperatively (Active Comparator): Patients undergoing laparoscopic inguinal hernia repair will stop Aspirin 5-7 days before the surgery
  Interventions: Procedure: Laparoscopic inguinal hernia repair without perioperative Aspirin
- Patients who continue Aspirin perioperatively (Experimental): Patients undergoing laparoscopic inguinal hernia repair will continue on Aspirin perioperatively
  Interventions: Procedure: Laparoscopic inguinal hernia repair with perioperative Aspirin

INTERVENTIONS:
Procedure: Laparoscopic inguinal hernia repair with perioperative Aspirin — Patients undergoing laparoscopic inguinal hernia repair will continue on Aspirin perioperatively
  Arms: Patients who continue Aspirin perioperatively
Procedure: Laparoscopic inguinal hernia repair without perioperative Aspirin — Patients undergoing laparoscopic inguinal hernia repair will stop Aspirin 5-7 days before the surgery
  Arms: Patients who stop Aspirin perioperatively

SUMMARY:
This study aims to assess the need to stop Aspirin before elective laparoscopic inguinal hernia repair. It will consist of 2 arms: patients who continue to take Aspirin perioperatively and patients who stop Aspirin 5-7 days before the surgery.

DETAILED DESCRIPTION:
This study aims to assess the need to stop Aspirin before elective laparoscopic inguinal hernia repair. It will consist of 2 arms: patients who continue to take Aspirin perioperatively and patients who stop Aspirin 5-7 days before the surgery. Simple randomization will be performed and allocation is via closed envelope method. The surgeon will be blinded regarding the usage of Aspirin. The primary outcome is the incidence of post-operative hematoma formation within the first 24 hours after surgery. The secondary outcomes are the incidence of post-operative seroma formation within 24 hours, the incidence of post-operative hematoma requiring intervention (including blood transfusion, percutaneous drainage and surgical hemostasis) within 30 days, pain at regular intervals and the incidence of other post-operative complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of inguinal hernia undergoing laparoscopic repair
* Age 21-80 years
* Patients taking Aspirin
* BMI 18-30

Exclusion Criteria:

* Age <21 and >80years
* Recurrent inguinal hernia
* Coagulopathy
* Patients who can't stop Aspirin
* BMI <18 and >30

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-04-01 (Actual); Primary Completion 2024-02-29 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of hematoma | 24 hours
  Postoperative scrotal or groin hematoma (not including skin bruising)

SECONDARY OUTCOMES:
Incidence of seroma | 24 hours
  Postoperative scrotal or groin seroma
Incidence of hematoma requiring intervention | 30 days
  Including blood transfusion, percutaneous drainage or surgical hemostasis

CONTACTS AND LOCATIONS:
Overall Officials: Davide Lomanto, MD PhD, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

REFERENCES:
- [Derived] Tan L, Yeow M, Fatt SLK, Parameswaran R, Mahipal M, Loo L, Wijerathne S, Lomanto D. Cessation vs no cessation of acetylsalicylic acid preoperatively in laparoscopic totally extraperitoneal inguinal hernia repair (CAPTAIN): final report from a multi-center, single-blinded, randomized-controlled trial. Hernia. 2025 Jul 5;29(1):221. doi: 10.1007/s10029-025-03418-4. PMID 40616699